CLINICAL TRIAL: NCT06164119
Title: A Randomised Effectiveness-implementation Trial for Evaluating Dietary and Manual Treatment With Osteopathic Techniques on Quality of Life and on Modulation of the Inflammatory State of Patients Diagnosed With Breast Cancer Undergoing Antiestrogenic Hormonal Treatment.
Brief Title: Effects of Diet and Osteopathy on Quality of Life and Inflammation in Breast Cancer Patients Under Hormonal Therapy
Acronym: SECCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: INT 107/23
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: hormonal therapy; treatment-related adverse events; osteopathic techniques; diet; quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an hybrid type I eﬀectiveness-implementation trial, testing the effectiveness of clinical therapeutic interventions, coupled by exploration of the eﬀects of the implementation of the effective intervention(s) in clinical practice (professional practice changes, changes in processes of care, quality of intervention delivery, patient's satisfaction).
  The effectiveness study will be a before-and-after randomized trial performed according to a 2 × 2 factorial design.
  Two groups are identified:
  * Group A: Premenopausal breast cancer patients treated with tamoxifen and/or luteinizing hormone-releasing hormone (LHRH) analogues.
  * Group B: Postmenopausal breast cancer patients treated with aromatase inhibitors.
  Patients in each group will be randomly assigned to four treatments arms:
  Arm 1, manual treatment with osteopathic techniques and nutritional treatment. Arm 2, manual treatment with osteopathic techniques. Arm 3, nutritional treatment. Arm 4, control.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- A1: manual treatment with osteopathic techniques and nutritional treatment in premenopausal patients (Experimental): Premenopausal breast cancer patients under tamoxifen and/or LHRH analogues are treated with manual treatment with osteopathic techniques (8 once-a-week manual treatments with osteopathic techniques) and nutritional treatment (personalized Mediterranean Diet).
  Interventions: Other: manual treatment with osteopathic techniques and nutritional treatment
- A2: manual treatment with osteopathic techniques in premenopausal patients (Experimental): Premenopausal breast cancer patients under tamoxifen and/or LHRH analogues are treated with manual treatment with osteopathic techniques (8 once-a-week manual treatments with osteopathic techniques).
  Interventions: Other: manual treatment with osteopathic techniques
- A3: nutritional treatment in premenopausal patients (Experimental): Premenopausal breast cancer patients under tamoxifen and/or LHRH analogues are treated with nutritional treatment (personalized Mediterranean Diet).
  Interventions: Other: nutritional treatment
- A4: control group in premenopausal patients (No Intervention): Premenopausal breast cancer patients under tamoxifen and/or LHRH analogues receive general counselling on healthy dietary habits and lifestyle in accordance to the World Cancer Research Fund (WCRF) guidelines.
- B1: osteopathic techniques and nutritional treatment in postmenopausal patients (Experimental): Postmenopausal breast cancer patients under aromatase inhibitors are treated with manual treatment (8 once-a-week manual treatments with osteopathic techniques) and nutritional treatment (personalized Mediterranean Diet).
  Interventions: Other: manual treatment with osteopathic techniques and nutritional treatment
- B2: manual treatment with osteopathic techniques in postmenopausal patients (Experimental): Postmenopausal breast cancer patients under aromatase inhibitors are treated with manual treatment with osteopathic techniques (8 once-a-week manual treatments with osteopathic techniques).
  Interventions: Other: manual treatment with osteopathic techniques
- B3: nutritional treatment in postmenopausal patients (Experimental): Postmenopausal breast cancer patients under aromatase inhibitors are treated with nutritional treatment (personalized Mediterranean Diet).
  Interventions: Other: nutritional treatment
- B4: control group in postmenopausal patients (No Intervention): Postmenopausal breast cancer patients under aromatase inhibitors receive general counselling on healthy dietary habits and lifestyle in accordance to the World Cancer Research Fund (WCRF) guidelines.

INTERVENTIONS:
Other: manual treatment with osteopathic techniques and nutritional treatment — manual treatment with osteopathic techniques (8 once-a-week manual treatments with osteopathic techniques) and nutritional treatment (personalized Mediterranean Diet)
  Arms: A1: manual treatment with osteopathic techniques and nutritional treatment in premenopausal patients; B1: osteopathic techniques and nutritional treatment in postmenopausal patients
Other: manual treatment with osteopathic techniques — manual treatment with osteopathic techniques (8 once-a-week manual treatments with osteopathic techniques)
  Arms: A2: manual treatment with osteopathic techniques in premenopausal patients; B2: manual treatment with osteopathic techniques in postmenopausal patients
Other: nutritional treatment — nutritional treatment (personalized Mediterranean Diet)
  Arms: A3: nutritional treatment in premenopausal patients; B3: nutritional treatment in postmenopausal patients

SUMMARY:
Breast cancer patients under hormonal therapy may experience significant adverse events related to this treatment and as a result, failure to adhere to adjuvant therapies or discontinuation of treatment has been reported to be high.

Promoting weight control and the adoption of healthy lifestyle habits in breast cancer survivors has an impact on hormonal status, quality of life and physical functioning, contributing to reduce cancer recurrence risk, cancer-related and chronic-condition-related mortality.

Manipulation procedures, such as manual treatment with osteopathic techniques, have positive effects on osteoarticular pain, peripheral neuropathies, anxious-depressive disorders, asthenia and sleep disorders, also improving immune and neuroendocrine responses.

The aim of this study is to evaluate the effects of dietary intervention and manual treatment with osteopathic techniques in women diagnosed with breast cancer under antiestrogenic hormonal treatment through the assessment of:

* modifications of quality of life (QoL)
* frequency and severity of symptoms related to antiestrogenic hormonal treatment
* body weight
* body composition
* food habits
* metabolic and inflammatory state
* physical performance
* patient's satisfaction to multidisciplinary treatment.

This study focuses on patient's centricity evaluating the effects that long lasting adjuvant therapies have on breast cancer survivors. Improving personalized patient's treatment through collaborative interactions between clinicians, osteopaths and nutrition specialists might result in implementation strategies to determine novel evidence-based treatments for ameliorating patient's adherence to oncological therapies, impacting prognosis and survival.

DETAILED DESCRIPTION:
Breast cancer patients under hormonal therapy may experience significant adverse events related to this treatment. Premenopausal women may encounter the classic symptoms of menopausal syndrome: hair thinning or loss; hot flashes, sweating, fatigue, insomnia, joint pain, vaginal dryness, decreased libido, anxious-depressive disorders, cognitive dysfunction; dry eyes; weight gain. Postmenopausal women may instead experience joint stiffness and joint pain, depressive and anxious symptoms, fatigue and irritability.

Since most of these adverse events do not resolve spontaneously a few weeks/months after starting treatment, they often negatively impact patient's quality of life.

As a result of treatment-related adverse events, failure to adhere to adjuvant therapies or discontinuation of treatment has been reported to be high and this may negatively impact patient's prognosis and survival.

Patients with breast cancer frequently experience weight gain during and after adjuvant hormonal treatment. Indeed, menopause, musculoskeletal pain and the consequent physical activity reduction, work together to reduce the basal energy metabolism. On the other side, the psychological distress and the eventual use of food for emotional reward, do promote weight gain. Notably, breast cancer patients who are overweight or obese show an increased risk of overall mortality, cancer-specific mortality, breast cancer relapse or second primary contralateral breast cancer. The explanation lies in the fact that the increase in fat mass is directly correlated to an increased production of estrogens, insulin, leptin and proinflammatory cytokines which, all together, exhibit a mitogenic activity on mammary cells. Proinflammatory cytokines and insulin deregulation on their turn, favor with time the onset of other chronic diseases such as diabetes, dyslipidemia, metabolic syndrome in general, thus increasing the risk of overall mortality. Conversely, weight loss can improve hormonal status, quality of life and physical functioning and contribute to reduce cancer recurrence risk, cancer-related and chronic-condition-related mortality. Therefore, it is important to promote weight control and the adoption of healthy lifestyle habits in breast cancer survivors.

Manipulation procedures, such as manual treatment with osteopathic techniques, involve the mechanical displacement of fluids and the removal of toxic substances with neurovascular and neuromuscular effects, thus producing positive alterations at the metabolic, biochemical and circulatory level. Several studies conducted on patients with breast cancer have supported the positive effect of manual therapy (acupuncture, shiatsu treatments, massages) on the control of various problems such as osteoarticular pain, peripheral neuropathies, anxious-depressive disorders, asthenia and sleep disorders, also improving immune and neuroendocrine responses.

Nevertheless, there are no studies on the effect of manual treatment with osteopathic techniques on the control of symptoms related to the side effects induced by anti-tumor therapies.

The aim of this study is to evaluate the effects of dietary intervention and manual treatment with osteopathic techniques in women diagnosed with breast cancer under antiestrogenic hormonal treatment through the assessment of:

* modifications of quality of life (QoL)
* frequency and severity of symptoms related to antiestrogenic hormonal treatment
* body weight
* body composition
* food habits
* metabolic and inflammatory state
* physical performance
* patient's satisfaction to multidisciplinary treatment.

This study focuses on patient's centricity evaluating the effects that long lasting adjuvant therapies have on breast cancer survivors. Improving personalized patient's treatment through collaborative interactions between clinicians, osteopaths and nutrition specialists might result in implementation strategies to determine novel evidence-based treatments for ameliorating patient's adherence to oncological therapies, impacting prognosis and survival.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Voluntary written informed consent
* Histologically confirmed estrogen receptor-positive invasive breast cancer or in situ breast cancer after breast surgery
* Absence of locoregional relapse or distant metastasis
* Premenopausal or postmenopausal status
* Hormonal therapy with tamoxifen and/or LHRH analogues or aromatase inhibitors
* Patients with or without neoadjuvant or adjuvant chemotherapy
* Patients with a BMI > 18.5 kg/m^2
* Absence of language barrier

Exclusion Criteria:

* Previous hormonal therapy
* Use of medical treatments that contrast adjuvant hormonal therapy adverse effects (e.g. menopausal symptoms and arthralgia).
* Underweight patients (BMI <18.5 kg/m^2)
* Patients diagnosed with eating disorders (e.g. anorexia nervosa, bulimia, binge eating, orthorexia)
* Psychiatric disorders or cognitive impairments
* Previous malignancies other than in situ cervical carcinoma or non-melanoma skin cancer
* Non-epithelial breast cancer at histological examination
* In situ lobular breast cancer
* Participation in other randomized clinical trials that could interfere with current study
* Patients living distant from trial center and unable to attend for check-ups and meetings.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effect of dietary intervention and manual treatment with osteopathic techniques on quality of life (QoL) of women diagnosed with breast cancer under hormonal treatment | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Quality of life will be assessed using the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) questionnaire comparing the before-and-after treatment difference in FACT-ES QoL scale (range 0-200; the higher the FACT-ES score, the better the quality of life, QoL) evaluated at baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3).
  The difference between pre treatment (baseline, T0) score and 24-weeks (six months, T2) score of the FACT ES QoL scale will be analyzed by ANOVA, and the interaction between the dietetic treatment and manual treatment with osteopathic techniques will be tested at 5% significance level. In a secondary ANOVA analysis, the baseline-to-52-weeks (T3) follow-up difference of the FACT ES QoL scale scores will additionally be analyzed.
  These analyses will be conducted separately in Groups A and B.

SECONDARY OUTCOMES:
Treatment-related adverse events of hormonal treatment in premenopausal and postmenopausal patients | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Symptoms related to hormonal treatment will be evaluated using Menopause Rating Scale (MRS) (range 0-44; higher scores indicating worse symptoms) in Group A and EORTC Quality of Life Questionnaire - Breast Cancer Module (EORTC-QLQ-C30/BR23) (range 0-100; higher scores corresponding to worse symptoms) in Group B, respectively.
Body weight | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Body weight will be evaluated using body mass index (BMI), measuring weight in kilograms divided by the square of height in meters.
Body composition | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Body composition will be evaluated combining two anthropometric measures: the waist circumference (cm) and calf circumference (cm).
Food habits | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Food habits will be assessed through a food frequency questionnaire.
Hemoglobin | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Hemoglobin will be assessed collecting blood exams measuring hemoglobin levels (g/dL).
Red blood cells | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Red blood cells will be assessed collecting blood exams measuring red blood cells count (cells/mcL).
Platelets | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Platelets will be assessed collecting blood exams measuring platelets count (cells/mcL).
White blood cells | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  White blood cells will be assessed collecting blood exams measuring white blood cells count (cells/mcL).
Lymphocytes | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Lymphocytes will be assessed collecting blood exams measuring lymphocytes count (cells/mcL).
Monocytes | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Monocytes will be assessed collecting blood exams measuring monocytes count (cells/mcL).
Neutrophils | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Neutrophils will be assessed collecting blood exams measuring neutrophils count (cells/mcL).
Inflammatory state: erythrocyte sedimentation rate | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  inflammatory state will be assessed collecting blood exams measuring erythrocyte sedimentation rate (ESR) (mm/h)
Vitamin D | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Vitamin D will be assessed collecting blood exams measuring Vitamin D levels (ng,mL).
Metabolic state: plasma glycemia | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Metabolic state will be assessed collecting blood exams measuring plasma glycemia (mg/dl)
Metabolic state: serum insulin concentration | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Metabolic state will be assessed collecting blood exams measuring serum insulin concentration (µU/ml).
Metabolic state: total cholesterol | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Metabolic state will be assessed collecting blood exams measuring total cholesterol (mg/dL).
Metabolic state: low-density lipoprotein (LDL) cholesterol | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Metabolic state will be assessed collecting blood exams measuring low-density lipoprotein (LDL) cholesterol (mg/dL).
Metabolic state: high-density lipoprotein (HDL) cholesterol | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Metabolic state will be assessed collecting blood exams measuring high-density lipoprotein (HDL) cholesterol (mg/dL).
Metabolic state: triglycerides | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Metabolic state will be assessed collecting blood exams measuring triglycerides (mg/dL).
Inflammatory state: c-reactive protein (CRP) | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  inflammatory state will be assessed collecting blood exams measuring c-reactive protein (CRP) (mg/L).
Sex hormone binding globulin (SHBG) | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Sex hormone binding globulin (SHBG) will be assessed collecting blood exams measuring sex hormone binding globulin levels (SHBG) (nmol/L).
Inflammatory state: Interleukin-6 (IL-6) | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  inflammatory state will be assessed collecting blood exams measuring Interleukin-6 (IL-6) levels (pg/mL).
Inflammatory state: Tumour necrosis factor-α (TNF-α) | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  inflammatory state will be assessed collecting blood exams measuring Tumour necrosis factor-α (TNF-α) levels (pg/ml).
Testosterone | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Testosterone levels will be assessed collecting blood exams measuring testosterone levels (ng/dL).
Modifications of blood lipid profile | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  modifications of blood lipid profile will be assessed collecting blood exams measuring plasma lipids by UPLC-MS.
Physical performance | baseline (T0), after 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Physical performance will be assessed using International Physical Activity Questionnaires (IPAQ) measuring physical activity levels (higher scores indicating higher physical activity).
Patient's satisfaction to multidisciplinary treatment | 12 weeks (T1), after 24 weeks (T2) and after 52 weeks (T3)
  Patient's satisfaction to multidisciplinary treatment will be assessed with Functional Assessment of Chronic Illness Therapy - Treatment Satisfaction - General questionnaire (FACIT-TS-G) (range 0-25; the higher the score, the better the satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Ferraris, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

REFERENCES:
- [Background] Sauter ER. Breast Cancer Prevention: Current Approaches and Future Directions. Eur J Breast Health. 2018 Apr 1;14(2):64-71. doi: 10.5152/ejbh.2018.3978. eCollection 2018 Apr. PMID 29774312
- [Background] Sharma R, Hamilton A, Beith J. LHRH agonists for adjuvant therapy of early breast cancer in premenopausal women. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD004562. doi: 10.1002/14651858.CD004562.pub3. PMID 18843661
- [Background] Martino G, Catalano A, Agostino RM, Bellone F, Morabito N, Lasco CG, Vicario CM, Schwarz P, Feldt-Rasmussen U. Quality of life and psychological functioning in postmenopausal women undergoing aromatase inhibitor treatment for early breast cancer. PLoS One. 2020 Mar 26;15(3):e0230681. doi: 10.1371/journal.pone.0230681. eCollection 2020. PMID 32214378
- [Background] Glaus A, Boehme Ch, Thurlimann B, Ruhstaller T, Hsu Schmitz SF, Morant R, Senn HJ, von Moos R. Fatigue and menopausal symptoms in women with breast cancer undergoing hormonal cancer treatment. Ann Oncol. 2006 May;17(5):801-6. doi: 10.1093/annonc/mdl030. Epub 2006 Feb 28. PMID 16507565
- [Background] Mantas, D., Kostakis, J.D. & Markopoulos, C. Aromatase inhibitors: A comprehensive review in mechanisms of action, side effects and treatment in postmenopausal early breast cancer patients. Hellenic J Surg 88, 245-251 (2016). https://doi.org/10.1007/s13126-016-0326-6
- [Background] Henry NL, Azzouz F, Desta Z, Li L, Nguyen AT, Lemler S, Hayden J, Tarpinian K, Yakim E, Flockhart DA, Stearns V, Hayes DF, Storniolo AM. Predictors of aromatase inhibitor discontinuation as a result of treatment-emergent symptoms in early-stage breast cancer. J Clin Oncol. 2012 Mar 20;30(9):936-42. doi: 10.1200/JCO.2011.38.0261. Epub 2012 Feb 13. PMID 22331951
- [Background] Sestak I, Cuzick J, Sapunar F, Eastell R, Forbes JF, Bianco AR, Buzdar AU; ATAC Trialists' Group. Risk factors for joint symptoms in patients enrolled in the ATAC trial: a retrospective, exploratory analysis. Lancet Oncol. 2008 Sep;9(9):866-72. doi: 10.1016/S1470-2045(08)70182-7. Epub 2008 Aug 12. PMID 18703382
- [Background] Vance V, Mourtzakis M, Hanning R. Relationships Between Weight Change and Physical and Psychological Distress in Early-Stage Breast Cancer Survivors. Cancer Nurs. 2019 May/Jun;42(3):E43-E50. doi: 10.1097/NCC.0000000000000612. PMID 29847347
- [Background] Kangas M, Henry JL, Bryant RA. Posttraumatic stress disorder following cancer. A conceptual and empirical review. Clin Psychol Rev. 2002 May;22(4):499-524. doi: 10.1016/s0272-7358(01)00118-0. PMID 12094509
- [Background] Kadakia KC, Snyder CF, Kidwell KM, Seewald NJ, Flockhart DA, Skaar TC, Desta Z, Rae JM, Otte JL, Carpenter JS, Storniolo AM, Hayes DF, Stearns V, Henry NL. Patient-Reported Outcomes and Early Discontinuation in Aromatase Inhibitor-Treated Postmenopausal Women With Early Stage Breast Cancer. Oncologist. 2016 May;21(5):539-46. doi: 10.1634/theoncologist.2015-0349. Epub 2016 Mar 23. PMID 27009936
- [Background] Murphy CC, Bartholomew LK, Carpentier MY, Bluethmann SM, Vernon SW. Adherence to adjuvant hormonal therapy among breast cancer survivors in clinical practice: a systematic review. Breast Cancer Res Treat. 2012 Jul;134(2):459-78. doi: 10.1007/s10549-012-2114-5. Epub 2012 Jun 12. PMID 22689091
- [Background] Hershman DL, Shao T, Kushi LH, Buono D, Tsai WY, Fehrenbacher L, Kwan M, Gomez SL, Neugut AI. Early discontinuation and non-adherence to adjuvant hormonal therapy are associated with increased mortality in women with breast cancer. Breast Cancer Res Treat. 2011 Apr;126(2):529-37. doi: 10.1007/s10549-010-1132-4. Epub 2010 Aug 28. PMID 20803066
- [Background] Greenlee H, DuPont-Reyes MJ, Balneaves LG, Carlson LE, Cohen MR, Deng G, Johnson JA, Mumber M, Seely D, Zick SM, Boyce LM, Tripathy D. Clinical practice guidelines on the evidence-based use of integrative therapies during and after breast cancer treatment. CA Cancer J Clin. 2017 May 6;67(3):194-232. doi: 10.3322/caac.21397. Epub 2017 Apr 24. PMID 28436999
- [Background] Hernandez-Reif M, Ironson G, Field T, Hurley J, Katz G, Diego M, Weiss S, Fletcher MA, Schanberg S, Kuhn C, Burman I. Breast cancer patients have improved immune and neuroendocrine functions following massage therapy. J Psychosom Res. 2004 Jul;57(1):45-52. doi: 10.1016/S0022-3999(03)00500-2. PMID 15256294
- [Background] Lissoni P, Messina G, Lissoni A, Franco R. The psychoneuroendocrine-immunotherapy of cancer: Historical evolution and clinical results. J Res Med Sci. 2017 Apr 26;22:45. doi: 10.4103/jrms.JRMS_255_16. eCollection 2017. PMID 28567065
- [Background] Borreani C, Alfieri S, Infante G, Miceli R, Mariani P, Bosisio M, Vernieri C, Bianchi GV, Capri G. Aromatase Inhibitors in Postmenopausal Women with Hormone Receptor-Positive Breast Cancer: Profiles of Psychological Symptoms and Quality of Life in Different Patient Clusters. Oncology. 2021;99(2):84-95. doi: 10.1159/000509651. Epub 2020 Sep 29. PMID 32992318
- [Background] Wolfenden L, Foy R, Presseau J, Grimshaw JM, Ivers NM, Powell BJ, Taljaard M, Wiggers J, Sutherland R, Nathan N, Williams CM, Kingsland M, Milat A, Hodder RK, Yoong SL. Designing and undertaking randomised implementation trials: guide for researchers. BMJ. 2021 Jan 18;372:m3721. doi: 10.1136/bmj.m3721. PMID 33461967
- [Background] Pearson N, Naylor PJ, Ashe MC, Fernandez M, Yoong SL, Wolfenden L. Guidance for conducting feasibility and pilot studies for implementation trials. Pilot Feasibility Stud. 2020 Oct 31;6(1):167. doi: 10.1186/s40814-020-00634-w. PMID 33292770
- [Background] Ingber DE, Wang N, Stamenovic D. Tensegrity, cellular biophysics, and the mechanics of living systems. Rep Prog Phys. 2014 Apr;77(4):046603. doi: 10.1088/0034-4885/77/4/046603. PMID 24695087
- [Background] Rizkalla MN, Henderson KK, Huntington-Alfano K, Heinking KP, Koronkiewicz A, Knees M, Hoffman H, Elahi F, Impens A. Does Osteopathic Manipulative Treatment Make a Neuropsychological Difference in Adults With Pain? A Rationale for a New Approach. J Am Osteopath Assoc. 2018 Sep 1;118(9):617-622. doi: 10.7556/jaoa.2018.136. PMID 30178052
- [Background] Williams NH, Hendry M, Lewis R, Russell I, Westmoreland A, Wilkinson C. Psychological response in spinal manipulation (PRISM): a systematic review of psychological outcomes in randomised controlled trials. Complement Ther Med. 2007 Dec;15(4):271-83. doi: 10.1016/j.ctim.2007.01.008. Epub 2007 Mar 8. PMID 18054729
- [Background] Vance V, Mourtzakis M, McCargar L, Hanning R. Weight gain in breast cancer survivors: prevalence, pattern and health consequences. Obes Rev. 2011 Apr;12(4):282-94. doi: 10.1111/j.1467-789X.2010.00805.x. Epub 2010 Sep 29. PMID 20880127
- [Background] Chan DSM, Vieira AR, Aune D, Bandera EV, Greenwood DC, McTiernan A, Navarro Rosenblatt D, Thune I, Vieira R, Norat T. Body mass index and survival in women with breast cancer-systematic literature review and meta-analysis of 82 follow-up studies. Ann Oncol. 2014 Oct;25(10):1901-1914. doi: 10.1093/annonc/mdu042. Epub 2014 Apr 27. PMID 24769692
- [Background] Majed B, Moreau T, Asselain B; Curie Institute Breast Cancer Group. Overweight, obesity and breast cancer prognosis: optimal body size indicator cut-points. Breast Cancer Res Treat. 2009 May;115(1):193-203. doi: 10.1007/s10549-008-0065-7. Epub 2008 Jun 12. PMID 18546073
- [Background] Rock CL, Byers TE, Colditz GA, Demark-Wahnefried W, Ganz PA, Wolin KY, Elias A, Krontiras H, Liu J, Naughton M, Pakiz B, Parker BA, Sedjo RL, Wyatt H; Exercise and Nutrition to Enhance Recovery and Good Health for You (ENERGY) Trial Group. Reducing breast cancer recurrence with weight loss, a vanguard trial: the Exercise and Nutrition to Enhance Recovery and Good Health for You (ENERGY) Trial. Contemp Clin Trials. 2013 Mar;34(2):282-95. doi: 10.1016/j.cct.2012.12.003. Epub 2012 Dec 22. PMID 23266440
- [Background] Patterson RE, Cadmus LA, Emond JA, Pierce JP. Physical activity, diet, adiposity and female breast cancer prognosis: a review of the epidemiologic literature. Maturitas. 2010 May;66(1):5-15. doi: 10.1016/j.maturitas.2010.01.004. Epub 2010 Jan 25. PMID 20097494
- [Background] Li CI, Daling JR, Porter PL, Tang MT, Malone KE. Relationship between potentially modifiable lifestyle factors and risk of second primary contralateral breast cancer among women diagnosed with estrogen receptor-positive invasive breast cancer. J Clin Oncol. 2009 Nov 10;27(32):5312-8. doi: 10.1200/JCO.2009.23.1597. Epub 2009 Sep 8. PMID 19738113
- [Background] Protani M, Coory M, Martin JH. Effect of obesity on survival of women with breast cancer: systematic review and meta-analysis. Breast Cancer Res Treat. 2010 Oct;123(3):627-35. doi: 10.1007/s10549-010-0990-0. Epub 2010 Jun 23. PMID 20571870
- [Background] Sauter ER, Scott S, Hewett J, Kliethermes B, Ruhlen RL, Basarakodu K, de la Torre R. Biomarkers associated with breast cancer are associated with obesity. Cancer Detect Prev. 2008;32(2):149-55. doi: 10.1016/j.cdp.2008.06.002. Epub 2008 Jul 17. PMID 18639389
- [Background] Hursting SD, Berger NA. Energy balance, host-related factors, and cancer progression. J Clin Oncol. 2010 Sep 10;28(26):4058-65. doi: 10.1200/JCO.2010.27.9935. Epub 2010 Aug 9. PMID 20697088
- [Background] Reeves MM, Terranova CO, Eakin EG, Demark-Wahnefried W. Weight loss intervention trials in women with breast cancer: a systematic review. Obes Rev. 2014 Sep;15(9):749-68. doi: 10.1111/obr.12190. Epub 2014 May 29. PMID 24891269
- [Background] Morey MC, Snyder DC, Sloane R, Cohen HJ, Peterson B, Hartman TJ, Miller P, Mitchell DC, Demark-Wahnefried W. Effects of home-based diet and exercise on functional outcomes among older, overweight long-term cancer survivors: RENEW: a randomized controlled trial. JAMA. 2009 May 13;301(18):1883-91. doi: 10.1001/jama.2009.643. PMID 19436015
- [Background] Newman AB, Simonsick EM, Naydeck BL, Boudreau RM, Kritchevsky SB, Nevitt MC, Pahor M, Satterfield S, Brach JS, Studenski SA, Harris TB. Association of long-distance corridor walk performance with mortality, cardiovascular disease, mobility limitation, and disability. JAMA. 2006 May 3;295(17):2018-26. doi: 10.1001/jama.295.17.2018. PMID 16670410
- [Background] Piccoli A, Rossi B, Pillon L, Bucciante G. A new method for monitoring body fluid variation by bioimpedance analysis: the RXc graph. Kidney Int. 1994 Aug;46(2):534-9. doi: 10.1038/ki.1994.305. No abstract available. PMID 7967368
- [Background] Buffa R, Mereu E, Comandini O, Ibanez ME, Marini E. Bioelectrical impedance vector analysis (BIVA) for the assessment of two-compartment body composition. Eur J Clin Nutr. 2014 Nov;68(11):1234-40. doi: 10.1038/ejcn.2014.170. Epub 2014 Aug 20. PMID 25139557
- [Background] Kim Y, Park I, Kang M. Convergent validity of the international physical activity questionnaire (IPAQ): meta-analysis. Public Health Nutr. 2013 Mar;16(3):440-52. doi: 10.1017/S1368980012002996. Epub 2012 Jul 2. PMID 22874087
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Bach-Faig A, Berry EM, Lairon D, Reguant J, Trichopoulou A, Dernini S, Medina FX, Battino M, Belahsen R, Miranda G, Serra-Majem L; Mediterranean Diet Foundation Expert Group. Mediterranean diet pyramid today. Science and cultural updates. Public Health Nutr. 2011 Dec;14(12A):2274-84. doi: 10.1017/S1368980011002515. PMID 22166184
- [Background] Vergnaud AC, Romaguera D, Peeters PH, van Gils CH, Chan DS, Romieu I, Freisling H, Ferrari P, Clavel-Chapelon F, Fagherazzi G, Dartois L, Li K, Tikk K, Bergmann MM, Boeing H, Tjonneland A, Olsen A, Overvad K, Dahm CC, Redondo ML, Agudo A, Sanchez MJ, Amiano P, Chirlaque MD, Ardanaz E, Khaw KT, Wareham NJ, Crowe F, Trichopoulou A, Orfanos P, Trichopoulos D, Masala G, Sieri S, Tumino R, Vineis P, Panico S, Bueno-de-Mesquita HB, Ros MM, May A, Wirfalt E, Sonestedt E, Johansson I, Hallmans G, Lund E, Weiderpass E, Parr CL, Riboli E, Norat T. Adherence to the World Cancer Research Fund/American Institute for Cancer Research guidelines and risk of death in Europe: results from the European Prospective Investigation into Nutrition and Cancer cohort study1,4. Am J Clin Nutr. 2013 May;97(5):1107-20. doi: 10.3945/ajcn.112.049569. Epub 2013 Apr 3. PMID 23553166
- [Background] Yumuk V, Tsigos C, Fried M, Schindler K, Busetto L, Micic D, Toplak H; Obesity Management Task Force of the European Association for the Study of Obesity. European Guidelines for Obesity Management in Adults. Obes Facts. 2015;8(6):402-24. doi: 10.1159/000442721. Epub 2015 Dec 5. PMID 26641646
- [Background] Lachenbruch PA. A note on sample size computation for testing interactions. Stat Med. 1988 Apr;7(4):467-9. doi: 10.1002/sim.4780070403. PMID 3368673
- [Background] FREEMAN GH, HALTON JH. Note on an exact treatment of contingency, goodness of fit and other problems of significance. Biometrika. 1951 Jun;38(1-2):141-9. No abstract available. PMID 14848119